CLINICAL TRIAL: NCT05985421
Title: Study of Gut Microbiota and Bacterial Translocation in Patients With Restless Legs Syndrome and Controls
Brief Title: Gut Microbiota and Bacterial Translocation in Restless Legs Syndrome
Acronym: RLS-BIOT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL23_0083
Record Dates: First submitted 2023-08-02; First posted 2023-08-14 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2023-08

CONDITIONS: Restless Legs Syndrome
Keywords: Periodic legs movement; Gut microbiota; Chronic inflammation; Iron metabolism
MeSH Terms: conditions — Restless Legs Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients
  Interventions: Other: Fecal collection; Other: Blood sampling; Other: Polysomnography; Other: Auto questionnaires
- Control
  Interventions: Other: Fecal collection; Other: Blood sampling; Other: Polysomnography; Other: Auto questionnaires

INTERVENTIONS:
Other: Fecal collection — approximate volume of 2 ml
Other: Blood sampling — 1 EDTA tube (7 ml) to test for chronic low-grade inflammation + 1 EDTA tube (7 ml) to test for intestinal inflammation, digestive permeability and microbial translocation
Other: Polysomnography — Polysomnography
Other: Auto questionnaires — International RLS Study Group Severity Scale, Epworth Sleepiness Scale, Insomnia Severity Index, Beck Depression Inventory-II, Autonomic symtoms scale (SCOPA-AUT)

SUMMARY:
Restless Legs Syndrome (RLS) is a common neurological sensorimotor disorder defined by an urge to move the legs when at rest that increase in the evening and at night. The pathophysiology of RLS remains poorly understood, but brain iron deficiency plays a major role. Iron absorption is an active process located in enterocytes of the proximal bowel, and is inhibited by hepcidin. The gut microbiota plays a central role in intestinal absorption, and in the maturation of the immune system. An imbalance in the microbiota, known as dysbiosis, could lead to a decrease in iron absorption, inflammation of the intestinal epithelium, and an increase in its permeability, thus favoring bacterial translocation and chronic systemic inflammation. Numerous studies showed an association between RLS and gastrointestinal diseases: Irritable bowel syndrome, Crohn's disease, ulcerative colitis, small intestinal bacterial overgrowth. However, no study has examined the gut microbiota in RLS.

The investigators hypothesize that there is an imbalance of gut microbiota in patients with RLS, favoring an increased intestinal permeability and bacterial translocation, leading to chronic inflammation and reduced iron bioavailability.

DETAILED DESCRIPTION:
Sixty patients with RLS will be included and 60 controls. The patients will be recruited from the active file of the sleep and wake disorders unit.

The control subjects will be recruited from :

* Patients hospitalized for suspected sleep disorders with normal PSG.
* The healthy controls of the RLS cognition protocol, ongoing in the department (ID-RCB: 2012-A00581-42, NCT01823354).

The patients will be informed of the study during a medical consultation. The consent of subjects participating in the study will be obtained during the pre-inclusion visit (D-1). The referring physician of the patients with RLS will propose them to participate in the study. After being duly informed of the nature, significance, implications of the study and appropriately documented by one of the investigators, and after sufficient time for reflection, free, informed and written consent will be obtained from all patients.

The control subjects will receive information about the study when they are admitted to hospital for polysomnographic recording, they will sign their consent for. A clinical examination will also be carried out.

ELIGIBILITY:
Inclusion Criteria:

Patient

* Idiopathic RLS diagnosed according to the 5 clinical criteria established by the IRLSSG (International Restless Legs Syndrome Study Group).
* Moderate to very severe RLS, IRLSSG questionnaire ≥ 15.
* Presence of periodic leg movements (PLM) during sleep (PLM index > 15/hour of sleep).
* Patient never treated or weaned at least 15 days prior to evaluation with dopaminergic agonists, alpha-2delta ligands, opioids or other psychotropic drugs.

Exclusion Criteria:

Patient

* Presence of digestive, inflammatory, psychiatric or neurological pathologies.
* C-reactive protein > 10mg/l (marker of acute inflammation)
* Presence of moderate-to-severe sleep apnea syndrome (apnea-hypopnea index >15/h).
* History of iron supplementation within 6 months.
* Use of treatments known to aggravate or cause RLS, such as antidepressants, neuroleptics, antihistamines or lithium.
* Refusal of consent after information
* legally protected adult (guardianship, curatorship)
* Pregnant or breast-feeding women
* Patient not affiliated to or not benefiting from a social security system.

Inclusion Criteria:

Control

* Adults without RLS with demographic characteristics similar to patients in terms of age (+- 5 years) and gender

Exclusion Criteria:

Control

* Presence of gastrointestinal, inflammatory, psychiatric or neurological diseases.
* C-reactive protein > 10mg/l (marker of acute inflammation).
* Presence of PLM in sleep (threshold >15 per hour of sleep).
* Treatment with antidepressants, neuroleptics, antihistamines, lithium, antiepileptics, benzodiazepines, hypnotics, opiates, dopaminergic agonists, levodopa, alpha-2delta ligands.
* Presence of moderate to severe sleep apnea syndrome (apnea-hypopnea index >15/h)
* Refusal of consent after information
* legally protected adult (guardianship, curatorship)
* Pregnant or breast-feeding woman
* Participant not affiliated to a social security scheme or not benefiting from such a system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 60 patients with RLS and 60 controls meeting all criteria, with the aim of having 50 analyzable subjects per group (i.e. with available stool samples).
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-01-09 (Actual); Primary Completion 2025-03-29 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Taxonomic composition of gut microbiota | 24 months
  Diversity (alpha and beta), abundance, nature and relative quantification of bacterial genera and bacterial taxonomic units (OTUs) present in stool samples identified by metagenomics.

SECONDARY OUTCOMES:
Ratio between Firmicutes and Bacteroidetes (majority phyla) | 24 months
  Richness, diversity and importance of minority phyla in stools, distribution and importance of bacterial genera in patients and controls. The study of the intestinal microbiota will consist of a metabarcoding approach to the V3-V4 regions of the 16S rRNA.

OTHER OUTCOMES:
Markers of intestinal inflammation (CD14s, LBP) | 24 months
  The study of bacterial translocation will be carried out using the ELISA technique for intestinal inflammation markers.
Markers of digestive permeability (I-FABP, claudine) | 24 months
  The study of bacterial translocation will be carried out using the ELISA technique for markers of membrane permeability.
Markers of microbial translocation (16S et 18SrDNA) | 24 months
  The study of bacterial translocation will be carried out using 16S and 18S qPCR for direct translocation markers.
Correspondence between bacteria identified by relative quantification of bacterial genera and OTUs present in stools and those detected by qPCR in plasma. | 24 months
  Identification of the concordance between bacterial genera identified in plasma and bacterial genera and OTUs present in stools will be done using Spearman's correlation coefficient.

CONTACTS AND LOCATIONS:
Overall Officials: DAUVILLIERS Yves, Pr, Principal Investigator — Head of Sleep/Wake Unit National reference center for orphan diseases Narcolepsy and hypersomnia
Locations (1):
- Unité des troubles du sommeil et de l'éveil-Centre de référence narcolepsie-Hypersomnie/Département de Neurologie/ Pole neurosciences tête et cou Hôpital Gui De Chauliac, Montpellier, France